CLINICAL TRIAL: NCT05796193
Title: Net Transition Initiative: Efficacy of Two Next-generation Nets for Control of Malaria in Cote D'Ivoire
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Institut Pierre Richet (Other Government); University of Ottawa (Other); University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28390
Record Dates: First submitted 2023-02-27; First posted 2023-04-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Malaria
Keywords: Anopheles density; Entomological inoculation rate; Malaria case incidence; Malaria infection prevalence
MeSH Terms: conditions — Malaria | interventions — cypermethrin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Py-PBO LLIN (Experimental): Veeralin is a long-lasting net of 130 deniers containing the pyrethroid insecticide alpha-cypermethrin 6.0 g/kg (216 mg/m2) and the synergist piperonyl butoxide (PBO) 2.2 g/kg (79.2 mg/m2) and manufactured by VKA polymers.
  Interventions: Other: Alpha-cypermethrin and PBO LLIN
- Py-CFP LLIN (Experimental): Interceptor® G2 is a long-lasting dual insecticide treated nets of 100 deniers combining Alpha-cypermethrin 2.4 g/kg (100 mg/m2) and Chlorfenapyr 4.8 g/kg (200 mg/m2) manufactured by BASF
  Interventions: Other: Alpha-cypermethrin and Clorfenapyr LLIN
- Py LLIN (Active Comparator): MAGNet® is a long-lasting net of 150 deniers containing the pyrethroid insecticide alpha-cypermethrin 5.8 g/kg (261 mg/m2) only and manufactured by VKA polymers.
  Interventions: Other: Alpha-cypermethrin only LLIN

INTERVENTIONS:
Other: Alpha-cypermethrin and PBO LLIN — Veeralin Long lasting insecticidal net with Alpha-cypermethrin Pyrethroid insecticide and PBO
  Arms: Py-PBO LLIN
Other: Alpha-cypermethrin and Clorfenapyr LLIN — Interceptor G2 dual active ingredient LLIN with with Alpha-cypermethrin Pyrethroid insecticide and Clorfenapyr
  Arms: Py-CFP LLIN
Other: Alpha-cypermethrin only LLIN — reference: standard pyrethroid LLIN
  Arms: Py LLIN

SUMMARY:
The investigator plan to conduct a three-arm cluster-randomized control trial which compares two next generation of long-lasting Insecticidal Nets (LLINs); Veeralin®LLIN (PBO-py LLIN), Interceptor G2 (chlorfenapyr-py LLIN) to a standard py-LLIN in the department of Tiebissou Southern Bouake city, central Côte d'Ivoire.

The primary objective of the project is to evaluate the efficacy of chlorfenapyr-pyrethroid and piperonyl-butoxide (PBO) synergist-pyrethroid LLINs on malaria case incidence in children aged 6 months to 10 years compared to standard pyrethroid-only LLINs. The secondary objectives are to evaluate the efficacy of the two intervention LLINs compared to the standard LLIN on a) malaria infection prevalence in the general population (both children and adults), b) vector density and c) entomological inoculation rate (EIR) (as a proxy for malaria transmission). In addition, changes in phenotypic resistance intensity and selection for molecular resistance mechanisms at baseline and 12 months post-LLIN distribution, in sentinel villages in each treatment arm will be investigate.

It is vital to demonstrate that these next generation LLINs which are becoming the standard of care in Sub Saharan AFRICA, are superior to standard py-LLIN in the most extreme resistance areas as this is likely where alternative interventions will be most needed to keep malaria control on track. The trial will generate the first epidemiological evidence on the efficacy of PBO nets compared to py-LLIN in West Africa.

DETAILED DESCRIPTION:
Background: The massive scale-up of long-lasting insecticidal nets (LLIN) has led to a major reduction in malaria burden in many sub-Saharan African (SSA) countries. This progress is threatened by the wide scale selection of insecticide resistant malaria vectors.

Study site: The study will be conducted in the department of Tiebissou (Gbeke Region in Lac district) Southern Bouake city, central Côte d'Ivoire. The Lac district is characterized by intense indoor malaria transmission with a prevalence of malaria reaching 51.3% in 2021 in children of under 5 years of age and extremely high pyrethroid resistance intensity in the main malaria vectors Anopheles gambiae s.s. and An. coluzzii.

Study design: Three-arm superiority, single blinded, cluster-randomised trial with village as the unit of randomisation. The arms consist of; 1/ Veeralin LLIN, a net combining the synergist PBO and the pyrethroid alpha-cypermethrin, 2/Interceptor G2, a mixture LLIN incorporating two adulticides with different modes of action; chlorfenapyr and a pyrethroid (alpha-cypermethrin), and 3/ the control arm: MAGNet LLIN, an alpha-cypermethrin-only LLIN.

Activities/Sample size:

A total of 33 villages (1 village = 1 cluster) with an average of 200 households will be identified and mapped. Nets will be distributed at a central point following national guidelines with 1 net for every 2 people.

To compare incidence of malaria cases between each intervention study arm and the control arm, a cohort of 50 children (45 + 5 to account for loss to follow up) will be recruited per cluster in 33 clusters for 12 months follow up to be able to detect a 35% relative reduction in malaria cases per child per year (rate ratio 0.65) between the intervention and the reference arms, assuming transmission in the control arm is 1.2 malaria cases per year with a coefficient of variation of 0.29 between clusters. The children will be visited twice a month during the transmission season (April to November) and once a month during the dry season.

Malaria infection prevalence cross-sectional surveys will be conducted, at baseline, 6 and 12 months after LLIN distribution. 50 people of all ages will be randomly selected from each of the 33 clusters (11 clusters per arm x 3 arms) and tested for malaria using RDT. The study will have 80% power to detect a relative 35% lower prevalence (prevalence ratio 0.65 in each intervention arm (VEERALLIN or Interceptor G2) relative to standard LLIN, assuming a prevalence of 50% in the control arm and a coefficient of variation of 0.3.

Vector density over 12 months will be followed using Human Landing Collection (HLC) indoor and outdoor with collection in 6 households in every cluster every 2 months. Assuming a mean mosquito density of 28 in the control arm, and a 60% reduction in mosquitoes in the intervention arms, with a coefficient of variation of 0.55 between clusters, this will give 80% power to detect differences at each timepoint.

Insecticide resistance intensity will be monitored at baseline and post intervention using adapted CDC bottle assays. The mechanism involved in resistance to pyrethroid and chlorfenapyr will be screened.

ELIGIBILITY:
Inclusion Criteria:

* For adults: willing to participate and provide consent
* For children: Having a parents/adult caregiver willing to provide written consent for the household and clinical survey and assent for children over 10
* Residing in the village over the last 3 months
* Be aged 6 months to 9 years old at time of recruitment (for the cohort)

Exclusion Criteria:

* Children who are expected to be non-resident over the period of study will be excluded (for the cohort)
* Dwelling not found or vacant during the survey (for prevalence and entomological surveys)
* No adult caregiver capable to give informed consent (All activities)
* Habitants/selected participants severely ill

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
malaria case incidence by malaria rapid diagnostic test HRP2/pLDH [pf/pan] | Over one year follow up
  Incidence of malaria cases (fever above 37.5C or history of a fever in the last 48 hours and a positive RDT) in children aged 6 months to 10 years.

SECONDARY OUTCOMES:
Malaria infection prevalence by malaria rapid diagnostic test HRP2/pLDH [pf/pan] | Baseline
  Malaria infection prevalence (by RDT) in the study population of all ages
Malaria infection prevalence by malaria rapid diagnostic test HRP2/pLDH [pf/pan] | 6 months post intervention
  Malaria infection prevalence (by RDT) in the study population of all ages
Malaria infection prevalence by malaria rapid diagnostic test HRP2/pLDH [pf/pan] | 12 months post intervention
  Malaria infection prevalence (by RDT) in the study population of all ages
Vector Density per person per night using human indoor and outdoor landing catches | Over one year follow up
  Indoor and outdoor Anopheles density per night per person
Sporozoite rate in Anopheles detected using Enzyme Linked Immuno-Sorbent Assay (ELISA) circumsporozoite protein technique. landing catches | Over one year follow up
  Proportion of Anopheles with malaria circumsporozoites in salivary gland
Mean number of Plasmodium spp infective malaria vectors collected per person per night | Over one year follow up
  Entomological inoculation rate measure as vector density x sporozoite rate

OTHER OUTCOMES:
gSG6-P1 IgG seroprevalence using ELISA technique | baseline
  Serological responses to mosquito salivary peptides: Blood spots on filter paper will be utilized to measure the level of antibodies in residents blood as a proxy for exposure to mosquito bites
gSG6-P1 IgG seroprevalence using ELISA technique | 12 months post intervention
  Serological responses to mosquito salivary peptides: Blood spots on filter paper will be utilized to measure the level of antibodies in residents blood as a proxy for exposure to mosquito bites
30 minutes mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | Baseline
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
24 hours mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | Baseline
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
72 hours mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | Baseline
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
30 minutes mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | 12 months post intervention
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
24 hours mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | 12 months post intervention
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
72 hours mortality in wild Anopheles post exposure to various concentration insecticide in CDC bottle assay | 12 months post intervention
  Phenotypic resistance to alpha-cypermethrin, PBO + alpha-cypermethrin and chlorfenapyr using WHO cylinder and CDC bottle bioassays will be conducted
Relative fold change in expression of metabolic genes | Baseline
  Selection for resistance will be monitored by measuring changes in levels of metabolic enzyme expression between wild population of Anopheles and susceptible reference Anopheles
Relative fold change in expression of metabolic genes | 12 months post intervention
  Selection for resistance will be monitored by measuring changes in levels of metabolic enzyme expression between wild population of Anopheles and susceptible reference Anopheles
Concentration of PBO, alpha-cypermethrin and Chlorfenapyr in g per kg in mosquito net | Before net distribution
  Concentration of chemical will be assessed by HPLC
24 hours and 72 hours mortality in a susceptible colony of Anopheles gambiae after exposure to new pieces of mosquito nets | Before net distribution
  Bio-efficacy testing will be conducted in standard WHO cone bio-assay and/or tunnel test
24 hours and 72 hours mortality in a resistant colony of Anopheles gambiae after exposure to new pieces of mosquito nets | Before net distribution
  Bio-efficacy testing will be conducted in standard WHO cone bio-assay and/or tunnel test

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Pierre Richet, Bouaké, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Sih C, Protopopoff N, Koffi AA, Ahoua Alou LP, Dangbenon E, Messenger LA, Kulkarni MA, Zoh MG, Camara S, Assi SB, N'Guessan R, Cook J. Efficacy of chlorfenapyr-pyrethroid and piperonyl butoxide-pyrethroid long-lasting insecticidal nets (LLINs) compared to pyrethroid-only LLINs for malaria control in Cote d'Ivoire: a three group, cluster randomised trial. Trials. 2024 Feb 28;25(1):151. doi: 10.1186/s13063-024-07969-2. PMID 38419075